CLINICAL TRIAL: NCT03501134
Title: ACTION: A Longitudinal Observational Study of Quality of Life, Functional Capacity and Physical Function in Glioblastoma Patients Treated With Tumor-Treating Fields
Brief Title: Quality of Life of Patients With Glioblastoma (GBM) Treated With Tumor-Treating Fields
Acronym: ACTION
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00088890
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Malignant Glioma
Keywords: Pro000888900; Katherine Peters; Optune; NovoTTF; ACTION; Quality of life; Tumor treating fields; Glioblastoma
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tumor treating fields: Patients diagnosed with WHO Grade IV malignant glioma who are approved and planned to use the NovoTTF device
  Interventions: Device: NovoTTF

INTERVENTIONS:
Device: NovoTTF — We are studying the effect of Tumor Treating Fields (NovoTTF), for example Optune™, on the quality of life, including exercise, sleep quality, and mood, of patients with malignant glioma who plan to use the NovoTTF device.

SUMMARY:
This purpose of this study is to describe the effect of Tumor Treating Fields (NovoTTF) on quality of life (QOL), including exercise, sleep quality, and mood, in patients with World Health Organization (WHO) Grade IV malignant glioma who have been prescribed and approved to receive Optune™. This is an observational, longitudinal study, meaning that information about QOL will be collected over time while the patient is using the NovoTTF device (for example, Optune™).

DETAILED DESCRIPTION:
Patients will be provided with a Fitbit Charge HR™, which they will begin wearing immediately to collect baseline information. The study team will teach the patients how to use the Fitbit and the associated smart phone application. Patients will also set an account with a platform that will provide information from the Fitbit (number of steps, sleep behaviors, and exercise log) to the study team. Patients will also have blood drawn, do a 6-minute walk test, and complete questionnaires at clinic visits 1, 8, 16, and 24 weeks after receiving the Fitbit. At the end of the study, patients will return the Fitbit to the study team.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to beginning specific protocol procedures
* Histologically proven World Health Organization (WHO) grade IV malignant glioma
* Completed standard-of-care treatment for newly diagnosed WHO grade IV malignant glioma, consisting of temozolomide (TMZ) and radiation therapy (RT)
* Signed Optune™ Prescription Form indicating intention of initiating NovoTTF therapy
* Stable disease status
* Patients ≥ 18 years of age
* Karnofsky Performance Status (KPS) ≥ 70
* Patient must be able to ambulate and complete the 6-minute walk test without use of a walker, cane, or any assist device
* Technology requirement:

  * Patients need to own a smart phone that can interface with the Fitbit Charge HR™.
  * Patients must be willing to provide their own internet access for this study. This will include either a data plan or Wi-Fi access on the patient's smart phone for use of the Fitbit Charge HR™ App. They will also need internet access (through their smart phone or home computer) for setting up a SGHIx account. Patients are welcome to use the free guest Wi-Fi access within the Duke Outpatient clinic area for the purpose of this study.
  * Patients will need a home computer or adaptor with USB port to charge the Fitbit Charge HR™.

Exclusion Criteria:

* Non-English speaking or inability to read and understand English.
* Presence of cardiovascular disease that would make physical activity risky, at the discretion of the provider.
* Any patient who is unable to comprehend and operate the activity tracker, at the discretion of the enrolling provider.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with WHO Grade IV malignant glioma who are approved for and intend to use NovoTTF therapy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Change in physical activity between baseline and week 24 | Baseline, 24 weeks
  Mean change between baseline and week 24 in total physical activity (MET-h/wk) as measured by the Godin Leisure Time Questionnaire

SECONDARY OUTCOMES:
Change in quality of life between baseline and week 24 | Baseline, 24 weeks
  Mean change from baseline at week 24 in subscales of the Functional Assessment of Cancer Therapy Brain (FACT-Br) and Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F)
Change in sleep quality between baseline and week 24 | Baseline, 24 weeks
  Mean change from baseline at week 24 in sleep quality as measured by the Pittsburgh Sleep Quality Assessment (PSQI)
Change in patient's mood state between baseline and week 24 | Baseline, 24 weeks
  Mean change from baseline at week 24 in mood as measured by the Beck Depression Inventory (BDI)
Change in functional capacity between baseline and week 24 | Baseline, 24 weeks
  Mean change from baseline at week 24 in functional capacity as measured by the 6-minute walk test
Change from baseline in average daily number of steps taken at 8, 16, and 24 (±3) weeks | Baseline, 8, 16, 24 weeks
  Mean change from baseline at week 8, 16, and 24 in the average daily number of steps as measured by the Fitbit among patients treated with Novo TTF

CONTACTS AND LOCATIONS:
Overall Officials: Katherine B Peters, MD, PhD, Principal Investigator — The Preston Robert Tisch Brain Tumor Center
Locations (1):
- The Preston Robert Tisch Brain Tumor Center at Duke, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — http://tischbraintumorcenter.duke.edu
- See also: Duke Cancer Institute — http://www.dukecancerinstitute.org/